CLINICAL TRIAL: NCT03264287
Title: Efficacy of Acupuncture Combined With Moving Cupping and Ear Point Tapping for Moderate and Severe Acne Vulgaris: A Randomized Controlled Trial
Brief Title: Efficacy of Acupuncture Combined With Moving Cupping and Ear Point Tapping for Moderate and Severe Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Chang Xie, Postgraduate student of Beijing University of Chinese Medicine & Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAMHospital20170301
Record Dates: First submitted 2017-08-09; First posted 2017-08-29 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; acupuncture; cupping; ear point tapping; randomized controlled trial
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 times per week therapeutic frequency (Experimental): 1.Acupuncture: GV20, LU5, LI11, LI4,GV14,BL13, ST2, BL2,ST7,ST6 and ashi point on the face.
  * Huatuo Brand needle (0.20*13mm) will be used for GV14, BL13, ST2, BL2, ST7, ST6 and ashi point on the face. Huatuo Brand needle (0.3*40mm) will be used for GV20, LU5, LI11 and LI4.
    2.Moving capping: Du Meridian (from GV14 to GV3) as well as the first (from BL11 to BL28) and second (from BL41 to BL53) side lines of the Urinary Bladder Meridian of Foot-Taiyang.
  * Guoyiyan Brand cupping jar (size 4) will be used. 3.Ear point tapping: Lung (CO14), Heart (CO15), Stomach (CO4), Neifenmi (CO18), Pizhixia (AT4).
  * Huatuo Brand, made by the seed of Vaccaria segetalis ( Neck.)Garcke.
  Interventions: Procedure: 3 times per week therapeutic frequency
- 1 time per week therapeutic frequency (Active Comparator): The acupoints and treating procedures will be the same as the 3 times per week group. Only treating frequency is different. The treating frequency is 1 time per week.
  1. Acupuncture: GV20, LU5, LI11, LI4,GV14,BL13, ST2, BL2,ST7,ST6 and ashi point on the face.
  2. Moving capping: Du Meridian (from GV14 to GV3) as well as the first (from BL11 to BL28) and second (from BL41 to BL53) side lines of the Urinary Bladder Meridian of Foot-Taiyang.
  3. Ear point tapping: Lung (CO14), Heart (CO15), Stomach (CO4), Neifenmi (CO18), Pizhixia (AT4).
     * Use the seed of Vaccaria segetalis ( Neck.)Garcke.
  Interventions: Procedure: 1 time per week therapeutic frequency

INTERVENTIONS:
Procedure: 3 times per week therapeutic frequency — Participants will receive acupuncture, moving cupping and ear-tapping procedure 3 times per week over the 6 weeks period.
  Arms: 3 times per week therapeutic frequency
Procedure: 1 time per week therapeutic frequency — Participants will receive acupuncture, moving cupping and ear-tapping procedure 1 time per week over the 6 weeks period.
  Arms: 1 time per week therapeutic frequency

SUMMARY:
This trial is designed to evaluate the efficacy of different frequencies in treating the moderate and severe acne vulgaris using acupuncture combined with moving cupping and ear point tapping.

DETAILED DESCRIPTION:
Background: Acne vulgaris is a common skin disease, especially in adolescents and young adults. Acne affects approximately 85% of teenagers, but can occur in most age groups and can persist into adulthood. There is no mortality associated with acne, but there is often significant physical and psychological morbidity. Acupuncture combined with moving cupping and ear point tapping may effectively relieve the skin lesions, but the evidence is limited. Also, young patients usually have no time to see the doctor frequently, thus it's necessary to figure out a better frequency of treating.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as acne vulgaris.
* GAGS score between 19 and 38 points.
* Age of 15 to 35 years.

Exclusion Criteria:

* Other types of acne: acne conglobate, acne fulminans，acne medicamentosa, premenstrual acne，cosmetic acne and trade acne.
* Presence of any other systemic disease that could affect the acne severity by its presence, such as polycystic ovarian syndrome, or thyroid diseases, or atypical congenital adrenal hyperplasia；or by any medication prescribed for the treatment of the systemic diseases.

  -- Use of any topical acne treatment or systemic antibiotics or traditional Chinese medicine within 2 weeks before study initiation. Use of a systemic retinoid within 9 months before study initiation. Use of a systemic steroid within 9 months before study initiation. Presence of any change in the use of oral contraceptive pills or anti-inflammatory drugs within 3 months before study initiation.
* Presence of any other skin disease that could interfere with the assessment of the acne, such as folliculitis or rosacea.
* Presence of severe heart, liver, kidney or hematopoietic system diseases, as well as severe malnutrition.
* Pregnancy or lactation.
* Recent use of this research scheme within 4 weeks before study initiation.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
IGA success rate | Baseline, week 1-6
  The proportion of subjects who achieved at least a two-point reduction from baseline to week 6 in IGA(Investigator's Global Assessment, scale from 0 to 5) score

SECONDARY OUTCOMES:
The change of IGA (Investigator's Global Assessment) score from baseline | Baseline, week 6, week 18, week 30
  After 6 weeks treating, the IGA(Investigator's Global Assessment, scale from 0 to 5) score's change from baseline.
The change of the Visual Analogue Scale (VAS) for facial pruritus from baseline | Baseline, week 6, week 18, week 30
  VAS uses a 100-mm line that is labeled at each end, and 0 mm represents no itch, and 100 mm represents unbearable itch. Patients will rate the VAS (average VAS of facial itch in the past 24 hours), and a researcher will record the VAS once weekly, generally at the third weekly treatment. The mean weekly VAS of itch over weeks 1-6 will be calculated as the sum VAS of each week divided by the number of weeks assessed.
The change of the Visual Analogue Scale (VAS) for facial lesion pain from baseline. | Baseline, week 6, week 18, week 30
  Visual Analogue Scale (VAS)VAS uses a 100-mm line that is labeled at each end, and 0 mm represents no pain, and 100 mm represents unbearable pain. Patients will rate the VAS (average VAS of facial pain in the past 24 hours), and a researcher will record the VAS once weekly, generally at the third weekly treatment. The mean weekly VAS of pain over weeks 1-6 will be calculated as the sum VAS of each week divided by the number of weeks assessed.
The change of the Total Lesion Count (TLC) on the face from baseline. | Baseline, week 6, week 18, week 30
  TLC is the sum of the inflammatory and non-inflammatory counts, including comedones, papules and pustules, nodules and cysts.
The change of the Inflammatory Lesions (IN) on the face from baseline. | Baseline, week 6, week 18, week 30
  IN is the sum of papules, pustules, nodules and cysts.
The change of the Skindex-16 dermatologic survey score from baseline. | Baseline, week 6, week 18, week 30
  Skindex-16 is a dermatologic quality-of-life survey. There are 16 questions in this survey. It concerns the skin condition which has bothered the patient the most during the past week. This survey calculated from 3 aspects including symptoms, emotions and functions. The score of each question is 0 to 6 points, and multiply by 16.6667，and get the sum of 16 questions' score. The average of the sum of 16 questions' score is the final result of skindex-16 dermatology survey. When the score is higher, it means the disease has greater influence on the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Song BH, Lee DH, Kim BC, Ku SH, Park EJ, Kwon IH, Kim KH, Kim KJ. Photodynamic therapy using chlorophyll-a in the treatment of acne vulgaris: a randomized, single-blind, split-face study. J Am Acad Dermatol. 2014 Oct;71(4):764-71. doi: 10.1016/j.jaad.2014.05.047. Epub 2014 Jun 12. PMID 24930587
- [Background] Zaenglein AL, Pathy AL, Schlosser BJ, Alikhan A, Baldwin HE, Berson DS, Bowe WP, Graber EM, Harper JC, Kang S, Keri JE, Leyden JJ, Reynolds RV, Silverberg NB, Stein Gold LF, Tollefson MM, Weiss JS, Dolan NC, Sagan AA, Stern M, Boyer KM, Bhushan R. Guidelines of care for the management of acne vulgaris. J Am Acad Dermatol. 2016 May;74(5):945-73.e33. doi: 10.1016/j.jaad.2015.12.037. Epub 2016 Feb 17. PMID 26897386
- [Background] Jung JY, Hong JS, Ahn CH, Yoon JY, Kwon HH, Suh DH. Prospective randomized controlled clinical and histopathological study of acne vulgaris treated with dual mode of quasi-long pulse and Q-switched 1064-nm Nd:YAG laser assisted with a topically applied carbon suspension. J Am Acad Dermatol. 2012 Apr;66(4):626-33. doi: 10.1016/j.jaad.2011.08.031. Epub 2011 Oct 26. PMID 22033354
- [Background] Eichenfield LF, Jarratt M, Schlessinger J, Kempers S, Manna V, Hwa J, Liu Y, Graeber M; Adapalene Lotion Study Group. Adapalene 0.1% lotion in the treatment of acne vulgaris: results from two placebo-controlled, multicenter, randomized double-blind, clinical studies. J Drugs Dermatol. 2010 Jun;9(6):639-46. PMID 20645525